CLINICAL TRIAL: NCT06121219
Title: Effect of Visual Retraining on Visual Loss Following Cortical Damage
Brief Title: Effect of Visual Retraining After Stroke
Acronym: urochester
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Krystel Huxlin, James V. Aquavella Professor of Ophthalmology, Associate Chair for Research, Dept. Ophthalmology, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008697
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Vision Loss Partial; Vision; Loss, Both Eyes; Hemianopia Homonymous; Hemianopia; Quadrantanopia; Stroke, Ischemic; Stroke - Occipital Infarction; Cortical Blindness
MeSH Terms: conditions — Blindness; Hemianopsia; Ischemic Stroke; Blindness, Cortical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Cortically Blind (CB) Subjects (Experimental): Cortically Blind subjects will be enrolled to perform a daily home visual training task.
  Interventions: Device: Training in the Blind Field
- Normative Comparator: Control Subjects (No Intervention): Healthy control subjects will be recruited to collect normative data by which to compare test results from CB subjects. No home training will be asked.

INTERVENTIONS:
Device: Training in the Blind Field — A computer software and chin-rest necessary to perform visual training will be loaned to each subject to be used at home. Subjects will perform one to two daily training sessions in their home, consisting of 200-300 trials each. The visual task performed repetitively will involve discriminating the direction of motion, the presence of motion, or the orientation of a visual stimulus (either a small cloud of dots or bars) located at a predetermined location in the blind field. The computer program will automatically create a record of patient performance during each home training session. Subjects will train daily (about 40-60 minutes total), 5 to 7 days per week for at least 3 and up to 12 months at a time.
  Arms: Experimental: Cortically Blind (CB) Subjects

SUMMARY:
This project is intended to collect data using standard clinical tests and psychophysics to quantify the effect of visual cortical damage on the structure of the residual visual system, visual perception, spatial awareness, and brain function. The investigators will also assess the effect of intensive visual retraining on the residual visual system, processing of visual information and the use of such information in real-world situations following damage. This research is intended to improve our understanding of the consequences of permanent visual system damage in humans, of methods that can be used to reverse visual loss, and of brain mechanisms by which visual recovery is achieved.

ELIGIBILITY:
Cortically Blind Subjects

Inclusion:

* Between 21 and 80 years of age
* Residents of the United States or Canada
* Unilateral stroke or stroke-like damage to primary visual cortex or its immediate afferent white matter sustained within the specified age range (21-75 years)
* Reliable visual field defects in both eyes as measured by Humphrey, MAIA, Goldmann, and/or equivalent perimetry, large enough to enclose a 5-deg diameter visual stimulus.
* Able to fixate on visual targets reliably for 1000ms
* Must have a home computer (desktop or laptop) and reliable internet access
* Willing, able, and competent to provide informed consent
* Normal cognitive abilities, able to understand written and oral instructions in English, and competent and responsible adults in order to complete the visual training at home, independently, as instructed, for several months.

Exclusion:

* Past or present eye disease interfering with visual acuity
* BCVA worse than 20/40 in either eye
* Damage to the dorsal Lateral Geniculate Nucleus
* Diffuse whole brain degenerative processes
* History of traumatic brain injury
* Any other brain damage deemed by study staff to potentially interfere with training ability or outcome measures
* Documented history of drug/alcohol abuse
* Currently taking neuroactive medications which would impact training, as determined by PI
* Presence of cognitive or seizure disorders
* One-sided attentional neglect
* Subjects who lack the competence or are otherwise unable to perform the visual training exercises as directed.

Control Subjects (n = 50)

Inclusion:

* Between 21 and 80 years of age
* Report no history of neurological disorder.
* Competent and responsible, as determined by the Principal Investigator.

Exclusion:

* Presence of damage to the visual system
* Presence of an active disease process involving their nervous system.
* Cognitive or seizure disorders
* Best corrected visual acuity worse than 20/40 in either eye
* Presence of vision field loss from ocular disease or disorder

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Direction Discrimination Threshold | Baseline to 4-6 months
  For each subject, the investigators will measure the change in ability to detect differences in the motion direction of visual stimuli relative to horizontal, measured in degrees of visual angle with respect to the stimulus. These assessments will be based on what can be reliably detected at a 72-75% correct level of performance on our 2AFC task, with task difficulty adjusted on a 3:1 staircase. The degrees of visual angle for the stimulus vary from 90 degrees (fully vertical) to 0.1 degrees (virtually overlapping the horizontal axis).
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training
Change in Mean Direction Discrimination Threshold | Baseline to 8-12 months
  For each subject, the investigators will measure the change in ability to detect differences in the motion direction of visual stimuli relative to horizontal, measured in degrees of visual angle with respect to the stimulus. These assessments will be based on what can be reliably detected at a 72-75% correct level of performance on our 2AFC task, with task difficulty adjusted on a 3:1 staircase. The degrees of visual angle for the stimulus vary from 90 degrees (fully vertical) to 0.1 degrees (virtually overlapping the horizontal axis).
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training
Change in Mean Direction Integration Threshold | Baseline to 4-6 months
  This will measure the change in ability of subjects to integrate across a range of motion directions measured in degrees of visual angle, with respect to the stimulus. These assessments will be based on what range of motion directions can be reliably integrated at a 72-75% correct level of performance on our 2AFC task, with task difficulty adjusted on a 3:1 staircase. The degrees of visual angle for the stimulus vary from 90 degrees (fully vertical) to 0.1 degrees (virtually overlapping the horizontal axis) .
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.
Change in Mean Direction Integration Threshold | Baseline to 8-12 months
  This will measure the change in ability of subjects to integrate across a range of motion directions measured in degrees of visual angle, with respect to the stimulus. These assessments will be based on what range of motion directions can be reliably integrated at a 72-75% correct level of performance on our 2AFC task, with task difficulty adjusted on a 3:1 staircase. The degrees of visual angle for the stimulus vary from 90 degrees (fully vertical) to 0.1 degrees (virtually overlapping the horizontal axis) .
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.
Change in Mean Contrast Sensitivity for Direction | Baseline to 4-6 months
  Assessment of visual perception transfer to untrained psychophysical tasks of contrast sensitivity for direction discrimination. This is a change metric as transfer must be compared from pre- to post- each course of training.
  For each subject, the investigators will measure the ability to correctly detect the motion direction of visual stimuli that are also varying in contrast against a grey background. The investigators will measure the luminance contrast, measured in percentage of contrast with respect to the stimulus, that can be reliably detected at a 72-75% correct level of performance. Contrast will vary between 100% (maximum contrast of black on grey) and 0.1% (minimum contrast visible of grey-on-grey) based on subject performance and a 3:1 staircase.
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.
Change in Mean Contrast Sensitivity for Direction | Baseline to 8-12 months
  Assessment of visual perception transfer to untrained psychophysical tasks of contrast sensitivity for direction discrimination. This is a change metric as transfer must be compared from pre- to post- each course of training.
  For each subject, the investigators will measure the ability to correctly detect the motion direction of visual stimuli that are also varying in contrast against a grey background. The investigators will measure the luminance contrast, measured in percentage of contrast with respect to the stimulus, that can be reliably detected at a 72-75% correct level of performance. Contrast will vary between 100% (maximum contrast of black on grey) and 0.1% (minimum contrast visible of grey-on-grey) based on subject performance and a 3:1 staircase.
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.
Change in Mean Contrast Sensitivity for Static Orientation | Baseline to 4-6 months
  Assessment of visual perception transfer to untrained psychophysical tasks of contrast sensitivity for static orientation discrimination. This is a change metric as transfer must be compared from pre- to post- each course of training.
  For each subject, the investigators will measure the ability to correctly detect the orientation of non-moving visual stimuli that vary in contrast against a grey background. The investigators will measure the luminance contrast, measured in percentage of contrast with respect to the stimulus, that can be reliably detected at a 72-75% correct level of performance. Contrast will vary between 100% (maximum contrast of black on grey) and 0.1% (minimum contrast visible of grey-on-grey) based on subject performance and a 3:1 staircase.
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.
Change in Mean Contrast Sensitivity for Static Orientation | Baseline to 8-12 months
  Assessment of visual perception transfer to untrained psychophysical tasks of contrast sensitivity for static orientation discrimination. This is a change metric as transfer must be compared from pre- to post- each course of training.
  For each subject, the investigators will measure the ability to correctly detect the orientation of non-moving visual stimuli that vary in contrast against a grey background. The investigators will measure the luminance contrast, measured in percentage of contrast with respect to the stimulus, that can be reliably detected at a 72-75% correct level of performance. Contrast will vary between 100% (maximum contrast of black on grey) and 0.1% (minimum contrast visible of grey-on-grey) based on subject performance and a 3:1 staircase.
  These measures of change will be evaluated baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.

SECONDARY OUTCOMES:
Humphrey 10-2 and 24-2 perimetry | Baseline to 4-6 months
  The investigators will measure the change in visual sensitivity (measured in decibels) at all locations tested by the system.
  These measures will be evaluated at baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.
Humphrey 10-2 and 24-2 perimetry | Baseline to 8-12 months
  The investigators will measure the change in visual sensitivity (measured in decibels) at all locations tested by the system.
  These measures will be evaluated at baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.
Goldmann perimetry | Baseline to 4-6 months
  The investigators will measure the change in area of vision (degrees squared) as encompassed by each isopter, measured by one of 3 different light stimuli.
  The 3 isopters which will be compared are:
  I2e 1asb, 0.25 mm^2 I4e 10asb, 0.25 mm^2 V4e 1000asb, 64 mm^2
  These measures will be evaluated at baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.
Goldmann perimetry | Baseline to 8-12 months
  The investigators will measure the change in area of vision (degrees squared) as encompassed by each isopter, measured by one of 3 different light stimuli.
  The 3 isopters which will be compared are:
  I2e 1asb, 0.25 mm^2 I4e 10asb, 0.25 mm^2 V4e 1000asb, 64 mm^2
  These measures will be evaluated at baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.
MAIA Visual Field Perimetry | Baseline to 4-6 months
  The investigators will measure the change in visual sensitivity (measured in decibels) at all locations tested by the system.
  These measures will be evaluated at baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.
MAIA Visual Field Perimetry | Baseline to 8-12 months
  The investigators will measure the change in visual sensitivity (measured in decibels) at all locations tested by the system.
  These measures will be evaluated at baseline and at each subsequent visit to the laboratory; minimally from baseline to 4-6 months, then baseline to 8-12 months from start of training.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No